CLINICAL TRIAL: NCT02585388
Title: A Randomized Phase II, Multicenter Study Evaluating the Benefit of Adding a Non Steroidal Aromatase Inhibitor to Oral Vinorelbine in Patients With Pretreated Metastatic Breast Cancer
Brief Title: Addition of Aromatase at the Navelbine in Pretreated Metastatic Breast Cancer.
Acronym: CHEOPS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Treatment toxicity
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-BR112
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
Keywords: pretreated metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Vinorelbine; Letrozole; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vinorelbine (Active Comparator): Vinorelbine (metronomic) alone 3 times per week ( mondays, wednesdays, Fridays or Thursdays, Tuesdays, Saturdays) at 50 mg per day, taken orally until progression of disease or toxicity.
  Interventions: Drug: Vinorelbine
- Vinorelbine+Anastrozole or Letrozole (Experimental): Vinorelbine metronomic 3 times per week (mondays, wednesdays, Fridays or Thursdays,Tuesdays, Saturdays) at 50 mg per day, taken orally until progression of disease or toxicity.
  And:
  Letrozole 2,5 mg every day or Anastrozole 1 mg every day. Until progression of disease or toxicity
  Interventions: Drug: Vinorelbine; Drug: Letrozole; Drug: Anastrozole

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine metronomic at 50 mg (1 tablet at 20 mg and 1 tablet at 30mg),per oral, 3 times per week. One dose level reduction is authorized at 30 mg per day.when stopping over 3 consecutive weeks due to toxicity, treatment should be permanently discontinued
  Other Names: Navelbine
Drug: Letrozole — Lestrozole at 2,5 mg every day , per oral
  Other Names: ARM A
  Arms: Vinorelbine+Anastrozole or Letrozole
Drug: Anastrozole — Anastrozole at 1 mg every day, per oral
  Other Names: ARM B
  Arms: Vinorelbine+Anastrozole or Letrozole

SUMMARY:
The CHEOPS study aims to confirm the clinical benefit of a combination of an anti-aromatase and metronomic chemotherapy treatment

DETAILED DESCRIPTION:
The CHEOPS study aims to confirm the clinical benefit of a combination of an anti-aromatase and metronomic chemotherapy treatment that would have the theoretical advantage of being well tolerated and more effective than chemotherapy alone even after an anti-aromatase therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 years.
2. Histologically proven breast cancer.
3. Progesterone and /or oestrogene receptors positive.
4. HER2 negative on primary tumour.
5. Patient taking hormonotherapy, in progression, already treated by at least one line of anti-aromatase non-steroidal hormonotherapy and by at least on line of chemotherapy.
6. Patient having to begin a second or third line of chemotherapy.
7. Presence of one or several measurable(s) or assessable(s) metastatic lesion(s).In case of isolated bone lesion (s): need to have a non-irradiated with an osteolytic component for be considered as lesion (s) target (s) and having an elevation of the CA15-3.
8. Post menopausal woman.
9. ECOG 0, 1 or 2.
10. Adequate biological function.

    * Neutrophil ≥ 1,5.E9/L
    * Platelets ≥ 100.E9/L
    * Creatinine clearance ≥ 30 mL/min
    * Total bilirubin ≤ 1,5 x the upper limit of normal (ULN)
    * Alkaline phosphatase ≤ 2,5 x ULN
    * ALT, AST ≤ 1,5 x ULN in the absence of liver metastases or ≤ 3 x ULN if liver metastases.
11. Patient with a life expectancy greater than 3 months.
12. Signed informed consent before enrollment.
13. affiliation to a social security scheme

Exclusion Criteria:

1. Patient with located or single metastatic tumoral relapse, accessible to a surgical treatment.
2. Patient having already received more 2 lines of chemotherapy for metastatic or advanced decease
3. Patient having already received a treatment by Navelbine®
4. Patient requiring an immediate located radiotherapy for analgesic action
5. Patient with non-irradiated cerebral or symptomatic metastasis, symptomatic pulmonary carcinomatosis lymphangitis
6. Simultaneous administration of another chemotherapy hormonotherapy or anti-tumoral drug
7. Patient having already received another treatment ongoing evaluation within the 30 days before the screening visit
8. Known positive serology HIV
9. Previous cancer within 5 years before the entry in the study, excepted an in situ carcinoma of the cervix or a spino or basal cell carcinoma of the skin or a nonmelanoma skin cancer with an adequate treatment.
10. Any serious concomitant pathology and / or uncontrolled could compromise participation in the study (including uncontrolled diabetes, uncontrolled hypertension, severe infection, profound malnutrition, unstable angina or congestive heart failure - class III or IV according to the New York Heart Association - ventricular arrhythmias, progressive coronary artery disease, myocardial infarction within the last six months, chronic liver or kidney disease, a progressive ulceration of the digestive tract above, CNS disorders).
11. Disorder of gastrointestinal function (GI) or pathology likely to significantly interfere with the absorption of Navelbine, of Letrozole or Anastrozole (eg. Ulcerative disease, uncontrolled nausea, vomiting, diarrhea, syndrome malabsorption, or resection of the small intestine).
12. Known hypersensitivity to letrozole, anastrozole, vinorelbine or other vinco-alkaloids or any other component.
13. Patient with fructose intolerance, galactose, a Lapp lactase deficiency or malabsorption of glucose and galactose (rare hereditary disease).
14. Patient with a history of poor compliance with medical treatment.
15. Patient can not be monitored regularly for family reasons, geographical, social or psychological.
16. Patient with altered mental status would not allow him to understand the study or give informed consent .

Ages: 50 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2017-05-15 (Actual); Study Completion 2017-05-15 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | up to 6 months
  Proportion of progression or death

SECONDARY OUTCOMES:
Evaluation of partial and complete response rate by RECIST 1.1 | up to 6 months
  partial and complete response rate by RECIST 1.1 in each arm
duration of response | up to 6 months
  duration of response is defined as the time from randomization and the disease progression
clinical benefit after 24 weeks of treatment | up to 24 weeks
  the clinical benefit is defined by the rate of complete response, by the rate of partial response and by the stability of lesions at 24 weeks according to criteria RECIST 1.1
overall survival | up to 2 years
  the overall survival of patients randomized is defined as the time from randomization and the date of death
Toxicity according to criteria NCI CTAEv4.03 | up to 2 years
  tolerance of the treatment based on AE occurrence according to criteria NCI CTAEv4.03
health-related quality of life | up to 2 years
  health-related quality of life and symptomatic state will be evaluated by filling a questionnaire by patients

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Etienne HEUDEL, MD, Principal Investigator — Centre Leon Berard
Locations (46):
- France (46):
  - Centre Hospitalier de l'Agglomération Montargoise, Amilly
  - ICO Paul Papin, Angers
  - Institut Sainte-Catherine, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - CHU de Brest, Brest
  - Clinique Pasteur, Brest
  - Centre Hospitalier Alpes Léman, Contamine-sur-Arve
  - CH de la Dracénie, Draguignan
  - Centre Hospitalier Intercommunal des Alpes du Sud, Gap
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - CHU de Grenoble, Grenoble
  - Hôpital Privé Drôme Ardèche - Clinique Pasteur, Guilherand-Granges
  - Hôpital Privé Drôme Ardèche, Guilhérand-Granges
  - CHD Vendée, La Roche-sur-Yon
  - Centre Hospitalier de Laon, Laon
  - CH Chartres Hôpital Louis Pasteur, Le Coudray
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Léon Berard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - CH Layne, Mont-de-Marsan
  - CH Montélimar, Montélimar
  - Centre Azuréen de Cancérologie, Mougins
  - Oracle, Nancy
  - Centre Catherine de Sienne, Nantes
  - CHR Orléans, Orléans
  - Centre Hospitalier de Pau, Pau
  - Polyclinique Francheville, Périgueux
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital privé des côtes d'armor, Plérin
  - Centre Hospitalier Annecy-Genevois, Pringy
  - Centre Hospitalier de la Région d'Annecy, Pringy
  - Centre Hospitalier de Quimper, Quimper
  - Institut du Cancer Courlancy Reims, Reims
  - Institut Jean Godinot, Reims
  - Centre Hospitalier de Romans sur Isère, Romans-sur-Isère
  - Hôpitaux Drôme Nord - Site de Romans, Romans-sur-Isère
  - CHP Saint Grégoire, Saint-Grégoire
  - ICO Gauducheau, Saint-Herblain
  - Polyclinique Côte Basque Sud, Saint-Jean-de-Luz
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Hospitalier de Soissons, Soissons
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpitaux du Léman, Thonon-les-Bains
  - Centre Hospitalier Jean Bernard, Valenciennes
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy